CLINICAL TRIAL: NCT06075654
Title: "Comparison of the Severity of Primary Dysmenorrhea Between Athletic and Non-Athletic Females: A Cross-Sectional Study" Comparison of the Severity of Primary Dysmenorrhea Between Athletic and Non-Athletic Females: A Cross-Sectional Study.
Brief Title: Primary Dysmenorrhea Severity in Athletic vs. Non-Athletic Females
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, khloud ramadan Abd El- fatah, principle investigator, Cairo University
Other Study IDs: P.T.REC/012/004091
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Primary Dysmenorrhea
MeSH Terms: interventions — Epidemiologic Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Athletic Group: athletic females complaining of primary dysmenorrhea, they participated in the exercise for the last ≥ 6 months, did exercises for ≥ 3 days/ week, and practiced (swimming, basketball, volleyball, gymnastics, judo, wrestling, karate, and boxing.
  Interventions: Other: no intervention it is considered (Epidemiological Study)
- Non-Athletic Group: Non-athletic females complaining form primary dysmenorrhea who are have not participated in any physical activity before
  Interventions: Other: no intervention it is considered (Epidemiological Study)

INTERVENTIONS:
Other: no intervention it is considered (Epidemiological Study) — It was a survey used Visual Analog Scale and WaLIDD scale to measure the severity of primary dysmenorrhea between both groups

SUMMARY:
The aim of the study is to investigate the difference in the severity of primary dysmenorrhea between athletic and non-athletic females.

DETAILED DESCRIPTION:
Primary dysmenorrhea is defined as colic pain in the lower abdomen which starts with the onset of menstruation. It is one of the most common gynecological disorders, an important cause of morbidity, and the most common cause of pelvic pain in menstruating girls and women it affects women in any age group. The prevalence varies widely, ranging from 17% to as high as 91%. Between 16% to 29% of women with dysmenorrhea have significant impairment in quality of life and the women's well-being. The rate of absenteeism from school, work, or other activities represents up to 15% of women with dysmenorrhea, dysmenorrhea is considered a source of considerable economic losses due to the costs of medications, medical care, and decreased productivity. Yoga, pilates, stretching, and other types of exercises have a noticeable effect on decreasing pain, and improving general health, and quality of sleep with different health conditions including primary dysmenorrhea. In addition, exercise and physical activity are used widely and proven to not only decrease pain but also improve quality of life, decrease stress, improve mental health, and in management of depression and stress.

For dysmenorrhea the mechanism that explained the effect of exercises on primary dysmenorrhea has been classified according to the intensity of the exercises; moderate -high-intensity exercise was believed to increase the anti-inflammatory cytokines, decrease the overall amount of prostaglandins released because of the decrease of the overall amount of menstrual flow. Low-intensity exercise reduces cortisol levels and prostaglandin synthesis

ELIGIBILITY:
Inclusion Criteria:

* Common inclusion criteria for athletic and non-athletic female.

  1. They had a regular menstrual cycle with a menstrual cycle length of 21-30 days.
  2. All females were virgins.
  3. Their ages ranged from 18 to 28 years old.
  4. Their BMI was ranged from 18.5 -29,9 kg/m2
  5. They did not use any pharmacological therapies for controlling pain during menstruation and during the application of the study.

Inclusion criteria athletic female:

1. They participated in the exercise for the last ≥ 6 months.
2. They did exercises for ≥ 3 days/ week.
3. They practiced (swimming, basketball, volleyball, ballet, gymnastics, judo, wrestling, karate, and boxing).

Exclusion Criteria:

1. History of pelvic pathology or any gynecological disease.
2. They had a history of chronic illness (eg: diabetes).
3. Their symptoms of dysmenorrhea became worse over time

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The athletic group will be selected from different clubs in Egypt for example; Benha, Tanta, Maadi, and Wadi-Degla clubs.
  Non- athletic will be selected from females and their their accompanying individuals
Sampling Method: Non-Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Data will be collected at a single time point, which is the baseline assessment
  The scale that will be used the VAS ;each subject will instructed to put point on line from no pain to tolerable pain

SECONDARY OUTCOMES:
Working ability, location, Intensity, Disability Dysmenorrhea scale. | Data will be collected at a single time point, which is the baseline assessment
  measuring a combination of manifestations: subjective (intensity /Wong-Baker, work ability) and objective (days of pain, location).
  In which each aspect of scale are rated from 0 to 3. 0 indicate no dysmenorrhea, 1-4 mild dysmenorrhea, 5-7 moderate dysmenorrhea, 8-12 sever dysmenorrhea.

CONTACTS AND LOCATIONS:
Locations (1):
- Khloud Ramadan Abd El- Fatah, Cairo, Egypt